CLINICAL TRIAL: NCT05978024
Title: Predicting Radiotherapy Response, Toxicities and Quality of Life Related Functional Outcome in Soft Tissue Sarcoma of the Extremities: a Prospective Observational Cohort Study
Brief Title: Predicting Radiotherapy Response and Toxicities in Soft Tissue Sarcoma of the Extremities - Cohort B
Acronym: PredicT-B
Status: Recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5166
Record Dates: First submitted 2023-07-14; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Soft Tissue Sarcoma of the Extremities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Tumour tissue for histopathological markers, immune function and DNA damage response from the area receiving radiotherapy (both biopsies and surgical resection specimens)
  * Blood samples for immune function analysis (Up to 50 ml at each time point).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicentre prospective cohort study, primarily aimed at reporting the frequency and intensity of radiotherapy side-effects of patients with soft tissues sarcoma of the extremities (STSE).

Two sub-studies are proposed within this study:

* MRI radiation response assessment Aimed at establishing whether changes in median apparent diffusion coefficients (ADC) are predictive of pre-operative STSE response measured using histopathology.
* Biomarker development and Immune mediators associated with radiotherapy Aimed at establishing prognostic markers which may refine selection of cases for pre-operative, palliative or no radiotherapy.

Also, aimed at determining if radiotherapy stimulates the tumour microenvironment, resulting in measurable change in anti-tumour immunity and if certain subtypes could potentially benefit from the addition of immunotherapy with radiation.

Patients participation in the sub-studies is optional.

DETAILED DESCRIPTION:
This is a multicentre prospective cohort study, primarily aimed at validating the dose-volume parameters identified in the analyses of the VorteX and IMRiS trials datasets.

• Delineation of healthy tissues

Pre-defined outlining guidelines of normal tissues as bones, muscle compartments, joints, lymph drainage basins and subcutaneous tissue from Predict A will be delineated in radiotherapy planning computed tomography (CT) images. All cases will be delineated by a single observer (Rita Simoes). Verification of all outlines will be carried out by Dr Aisha Miah (clinical supervisor).

• Dose-volume constraints validity testing

Patients will be treated as per local protocol treatment technique.

Radiotherapy, clinical and toxicities data will be collected, with no new intervention on the treatment. Patients enrolled will receive standard radiation prescription doses as described below:

* Pre-operative radiotherapy- 50 Gy in 25 fractions equivalent (pre-operative radiotherapy). Where appropriate hypo-fractionated schedules as per institutional guidelines can considered: eg. 25 Gy/ 5 daily fractions. In myxoid liposarcomas, 36 Gy in 18 fractions can be considered where suitable;
* Post-operative radiotherapy- 60 Gy in 30 fractions or 66 Gy in 33 fractions (positive resection margins); alternative hypo-fractionated schedules as per institutional guidelines can be considered;
* Palliative radiotherapy- 30-36 Gy in 10-12 daily fractions, 40-45 Gy in 15 fractions, 30-36 Gy in 5-6 once weekly fractions or 25 Gy in 5 daily fractions.

Toxicity will be assessed with the TESS and RTOG scoring instruments and Stern score for lymphoedema. Patients enrolled in the study will fill in a specific quality-of-life questionnaire to assess quality of life related functional outcomes following treatment for STSE. This questionnaire is based on validated questions for assessing quality-of-life. Patients will be followed up at 3, 6, 12, 18, and 24 months post-radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological diagnosis of soft tissue sarcoma of the upper or lower limb or limb girdle;
* Patients receiving pre-operative (neo-adjuvant), post-operative (adjuvant) or palliative radiotherapy;
* Patients receiving radiotherapy planned as per local protocols (neoadjuvant chemotherapy will be allowed). Neoadjuvant chemotherapy patients may be approached as they commence chemotherapy;
* WHO performance status 0-2;
* Aged ≥16 years;
* Patients fit enough to undergo radiotherapy treatment and willing to attend follow up visits, during two years;
* Female patients of child-bearing potential and male patients with partners of child-bearing potential must agree to use adequate contraception methods, which must be continued for 3 months after completion of treatment;
* Capable of giving written informed consent.

Exclusion Criteria:

* Previous radiotherapy to the same site;
* Pregnancy;
* Patients with concurrent or previous malignancy that could compromise assessment of primary and secondary endpoints of the trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population to be enrolled in this observational study will have had been diagnosed with STSE and referred to receive a course of radiotherapy either in the primary, palliative, pre-operative or post-operative settings.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of any RTOG grade ≥ 2 toxicities following treatment for STSE at 24 months | 24 Months
  The primary objective is to report the frequency and intensity of radiotherapy side-effects in STSE.

SECONDARY OUTCOMES:
The ability of the fitted model from dose-volume constraints from PredicT A (IMRiS and Vortex analysis) to correctly predict the incidence of grade 2+ among PredicT B patients. | 24 Months
  To report the differences in experienced by patients with STSE for whom dose-volume constraints were below or exceeded. Binary logistic regression will be used to quantify the differences using odds ratios (OR) from the fitted models. Univariate logistic regression models will be fitted to predict for the parameters relevant to toxicity grades in the RTOG, Stern's and TESS scales. ORs for each of the parameters will be used to judge for significant differences between the groups. There is no plan to fit multivariate model.
To report frequencies and proportions of radiotherapy-induced late toxicities | 24 Months
  Frequencies and proportions of radiotherapy-induced late toxicities at the specified at 3, 6, 12, 18 and 24 months will be reported descriptively at each time point for the overall events and by types of events:
  1. Subcutaneous tissue fibrosis
  2. Lymphoedema
  3. Bone fractures
  4. Joint stiffness
  5. Delayed wound healing following pre-operative RT
To determine the time to developing early and late side-effects. | 24 Months
  Time elapsed between day 1 of radiotherapy and the day to develop early and late side-effects using Kaplan-Meier methods. Median time to early side-effects with 95% confidence interval will be reported. Patients without any side-effects (on day 90 from end of RT) will be censored. Similarly, median time to late side-effects with 95% confidence interval will be reported. Patients without an event will be censored at the 24 months assessment visit or at last follow-up date known to be on the study without any event.
To determine radiological response rates to radiotherapy and where applicable chemo-radiotherapy for STSE of different histological subtypes. | 24 Months
  Differences in the tumour volumes (in cc and %) will be calculated from CT and CBCT images at fractions 8, 16 and 25 for patients receiving pre-operative RT. Changes in target volumes during radiotherapy will be assessed by computing dissimilarity indices (e.g., Simpson's dissimilarity index) in sequential CBCT images captured during treatment compared to radiotherapy planning CT. Radiological: % volume change (RECIST), % cystic sold component).
To determine histological response rates to radiotherapy and where applicable chemo-radiotherapy for STSE of different histological subtypes. | 24 Months
  Differences in the response rates will be assessed according to: histopathological semi-quantitative scores (pathological: % viable cells). Tumour factors are tumour histotype, staging and tumour size.
To determine quality of life-related functional outcomes and explore correlations with dose-volume parameters for patients who have received pre, post-operative or palliative radiotherapy for STSE. | 24 Months
  Correlations between functional outcomes (expressed in TESS and EORT-QLQ- C30 and QLQ-FA12 fatigue questionnaire scores) with dose-volume parameters (expressed in Gy/volume, where volume will be defined in % of total volume and cc) will be calculated using Spearman's correlation method. Patients will be categorised according to dose volume constraints and compare the groups using t-test or Mann-Whitney non-parametric test as appropriate.
To determine predictive and prognostic factors for local and distant recurrence and overall survival for patients receiving pre-operative and palliative RT. | 24 Months
  Percentage of patients responding to treatment will be calculated, this will be reported in the overall patients and for dose-volume constraints groups. Local control rates, disease-free survival rates and overall survival at 2 years will be calculated using Kaplan-Meier methods. Disease free survival events are local or distance disease recurrence and death from disease related causes. Overall survival events are death from any causes.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Miah, Principal Investigator — The Royal Marsden Hospital
Locations (3):
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge
  - The Royal Marsden NHS Foundation Trust, London
  - University College London, London

IPD SHARING:
Plan to Share IPD: No
Patient outcomes data will be utilised to publish study endpoints. However specific participant data will not be shared.
  We aim to publish protocol, and study results in the form of peer-reviewed publications and guidelines

REFERENCES:
- [Derived] Simoes R, Gulliford S, Seddon B, Dehbi HM, Robinson M, Forsyth S, Hughes A, Gaunt P, Nguyen TG, Elston S, Mohammed K, Zaidi S, Miles E, Hoskin P, Harrington K, Miah A. Predicting radiotherapy response, Toxicities and quality-of-life related functional outcomes in soft tissue sarcoma of the extremities (PredicT) using dose-volume constraints development: a study protocol. BMJ Open. 2024 Aug 9;14(8):e083617. doi: 10.1136/bmjopen-2023-083617. PMID 39122389